CLINICAL TRIAL: NCT03926793
Title: A Phase 1b, Randomized, Subject- and Investigator-Blinded, Placebo-Controlled, Multi-Center Clinical Trial to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Biomarkers of Inhaled GB002 in Subjects With WHO Group 1 Pulmonary Arterial Hypertension (PAH)
Brief Title: Clinical Study of Inhaled GB002 for Treatment of WHO Group I Pulmonary Arterial Hypertension
Acronym: PAH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GB002, Inc., a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GB002-1101
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Clinical site investigators, study personnel, and study subjects will be blinded to treatment assignment; however, the Sponsor will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Cohort 1 (Experimental): Patients will be randomized to receive inhaled GB002 or Placebo daily for 14 days
  Interventions: Drug: GB002; Drug: Placebo; Device: Generic Dry Powder Inhaler
- Cohort 2 (Experimental): Patients will be randomized to receive inhaled GB002 or Placebo daily for 14 days
  Interventions: Drug: GB002; Drug: Placebo; Device: Generic Dry Powder Inhaler
- Open Label Extension (Experimental): Eligible subjects may participate in the Open Label Extension (OLE) study for a period of 24 weeks.
  Interventions: Drug: GB002; Device: Generic Dry Powder Inhaler

INTERVENTIONS:
Drug: GB002 — GB002 low dose or high dose for inhalation
Drug: Placebo — Placebo for inhalation
  Arms: Cohort 1; Cohort 2
Device: Generic Dry Powder Inhaler — Generic dry powder inhaler for GB002 or Placebo delivery

SUMMARY:
This is a Phase 1B, randomized, participant- and investigator-blinded, placebo-controlled, multi-center clinical trial to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and biomarkers of inhaled GB002 in adults with World Health Organization (WHO) Group 1 Pulmonary Arterial Hypertension (PAH).

DETAILED DESCRIPTION:
The primary objective for this trial is to evaluate the safety and tolerability of GB002. The secondary objective for this trial is to evaluate the PK parameters of GB002. Exploratory objectives are to evaluate the PD readouts, change in WHO Group I functional class, and change in quality of life associated with GB002 treatment.

In this Phase 1B study, two dose levels of GB002 will be tested in adult participants with PAH. Four participants in cohort 1 will be randomized to receive up to two daily doses of either active drug or placebo, with 3 subjects receiving GB002 and 1 subject receiving placebo. An additional 4 participants (3 active and 1 placebo) may be added to cohort 1 at the discretion of the Data Review Committee (DRC). The dose and dosing interval (i.e., once daily or twice daily) for the second cohort will be determined by review of the safety, tolerability, and drug levels in the blood from cohort 1. Cohort 2 participants will also be randomized such that 6 subjects receive GB002 and 2 subjects receive placebo.

Eligible subjects who have completed the 2 week treatment period have the option to participate in a 24 week open label extension.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (males and females) aged 18 to 75 years (inclusive) with pulmonary arterial hypertension (PAH) (Main study)
2. A current diagnosis of symptomatic PAH classified by one of the following (Main and OLE study):

   1. Idiopathic (IPAH) or heritable pulmonary arterial hypertension (HPAH)
   2. PAH associated with one of the following connective tissue diseases (CTDs):

      systemic sclerosis, rheumatoid arthritis, mixed CTD or overlap syndrome, or systemic lupus erythematosus
   3. PAH associated with anorexigen or methamphetamine use
3. World Health Organization (WHO)/New York Heart Association (NYHA) functional class II-IV symptomatology (Main study)

Exclusion Criteria:

1. Clinically significant systemic hypertension or hypotension (Main and OLE study)
2. History of left-sided heart disease and/or clinically significant cardiac disease (Main and OLE study)
3. History of decompensated right heart failure within 30 days of screening (e.g., hospitalization for PAH or the need to add an additional PAH medication) (Main study)

NOTE: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Related Adverse Events GB002 (Main study) | Up to 45 days
  To evaluate the safety and tolerability of GB002
Number of participants with Treatment-Related Adverse Events GB002 (OLE study) | Up to 200 days
  To evaluate the long-term safety and tolerability and efficacy of GB002

SECONDARY OUTCOMES:
Pharmacokinetics: Time to Reach Maximum Concentration (Tmax) of GB002 (Main study) | 14 days
Pharmacokinetics: Maximum Concentration (Cmax) of GB002 (Main study) | 14 days
Pharmacokinetics: Area Under the Concentration Curve (AUC) of GB002 (Main study) | 14 days
Changes from baseline in 6-Minute Walk Test (6MWT) (OLE study) | 169 days
Changes from baseline in WHO Functional Class (OLE study) | 197 days
Changes from baseline in N-terminal pro B-type natriuretic peptide (NT-proBNP) (OLE study) | 169 days
Changes from baseline in Pulmonary Arterial Hypertension - Symptoms and Impact (PAH-SYMPACT) Quality of Life questionnaire (OLE study) | 197 days
Changes from baseline in Right Ventricular function by imaging (OLE study) | 169 days

CONTACTS AND LOCATIONS:
Locations (14):
- United States (12):
  - UCSD Medical Center, La Jolla, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Duke Early Phase Research, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center Montefiore University Hospital, Pittsburgh, Pennsylvania
  - VitaLink Research - Anderson, Anderson, South Carolina
- United Kingdom (2):
  - Golden Jubilee National Hospital, Glasgow
  - Hammersmith Hospital, Imperial Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No